CLINICAL TRIAL: NCT02465658
Title: Risk Factors for Co-existence of Cervical Elongation in Uterine Prolapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503073RIND
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: uterine prolapse; cervical elongation; pelvic floor reconstruction surgery
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Medical records were reviewed. — retrospective study

SUMMARY:
The presence of co-existence of cervical elongation in women of uterine prolapse may decrease the patients' satisfaction of uterine-preservation surgery for uterine prolapse, and additional surgery, such as Manchester surgery, may be needed to solve the problem.Thus the aim of this study is to investigate the risk factors of co-existence of cervical elongation in uterine prolapse.

DETAILED DESCRIPTION:
Purpose:

Thus the aim of this study is to investigate the risk factors of co-existence of cervical elongation in uterine prolapse.

Patients and Methods:

Between January 1994 and October 2014, all women underwent vaginal total hysterectomy in a medical center were enrolled in this study. Medical records were reviewed. Cervical elongation is defined as the presence of cervical length >3.38 cm or cervix to corpus ratio >0.79.

Expected Results:

The investigators will get the risk factors of co-existence of cervical elongation in uterine prolapse, and the result should be helpful for preoperative consultation, especially for uterine-preserving pelvic floor reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* All women with uterine prolapse underwent vaginal total hysterectomy
* > 20 years old.

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with uterine prolapse and underwent vaginal total hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Factors associated with coexistent cervical elongation in cases with uterine prolapse | 1 day
  Medical record review

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynecology, National Taiwan University Hospital, Taipei, Taiwan, Taiwan